CLINICAL TRIAL: NCT02969707
Title: Use of Repetitive Transcranial Magnetic Stimulation to Augment Hypnotic Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David Spiegel, Willson Professor and Associate Chair of Psychiatry & Behavioral Sciences, Director of the Center on Stress and Health, and Medical Director of the Center for Integrative Medicine at Stanford University School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 38138; 1R33AT009305-01 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Results first posted 2021-08-30 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
Keywords: repetitive Transcranial Magnetic Stimulation; functional MRI; Fibromyalgia; Hypnosis; Pain Assessment
MeSH Terms: conditions — Fibromyalgia | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind sham vs. real rTMS; data analysts blind to group assignment; subjects debriefed on their guess about sham vs. real - no better than chance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active rTMS (Experimental): The active group will receive repetitive Transcranial Magnetic Stimulation
  Interventions: Device: MagPro TMS system (MagVenture, Denmark); Behavioral: Hypnosis
- Sham rTMS (Sham Comparator): The sham repetitive Transcranial Magnetic Stimulation group will have the stimulation blocked.
  Interventions: Device: MagPro TMS system (MagVenture, Denmark); Behavioral: Hypnosis

INTERVENTIONS:
Device: MagPro TMS system (MagVenture, Denmark) — The investigators will perform two applications of 40s of continuous theta-burst stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left DLPFC will be determined by Localite Neuronavigation and targeted at the posterior middle frontal gyrus. The baseline structural scan obtained during the scan 1 will be utilized for this localization process. rTMS will be delivered using a MagPro TMS system (MagVenture, Denmark). sham rTMS will be delivered using a MagPro TMS system (MagVenture, Denmark).sham rTMS will be delivered using a MagPro TMS system (MagVenture, Denmark).
  Other Names: rTMS will be delivered using the MagPro TMS system (MagVenture, Denmark).
Behavioral: Hypnosis — Hypnotizability will be measured using the Hypnotic Induction Profile before and after administration of real vs. sham rTMS. Hypnotizability will be measured using the Hypnotic Induction Profile before and after administration of real vs. sham rTMS. Hypnosis will be employed to influence Stroop performance (conflict detection) and for pain management. The hypnotic instructions for this will be pre-recorded and played during fMRI.

SUMMARY:
The investigators plan to use functional neuroimaging (fMRI) to understand the brain systems affected when hypnosis and hypnotic analgesia are augmented with repetitive transcranial magnetic stimulation (rTMS), a form of non-invasive brain stimulation to 100 people with fibromyalgia, a chronic pain condition. The investigators will measure the effect of rTMS-augmentation on the brain networks underlying hypnotizability, as well as the effect of rTMS-augmentation on hypnotic analgesia networks. The investigators hope to demonstrate that a combination of these psychological and neuromodulatory treatments will be more effective than hypnosis alone, thereby enhancing the depth of hypnosis, range of hypnosis and the efficacy of hypnotic analgesia and hopefully creating a new treatment modality for individuals suffering from pain syndromes such as fibromyalgia pain.

DETAILED DESCRIPTION:
Overall Study Design. The investigators propose to develop a combinatory approach where an integrative technique (hypnosis) is augmented with a neurotechnology (repetitive transcranial magnetic stimulation). This application seeks to utilize the previously established brain-based mechanisms of both hypnosis and repetitive transcranial magnetic stimulation as biomarkers to assess the potential synergistic mechanism of this combinatory approach. 100 low-moderately hypnotizable subjects with fibromyalgia will be identified. The subjects' response to rTMS-augmentation of hypnosis will be measured. The volunteers will be randomized to active or sham rTMS. Two scan sessions will be performed for each subject, with the first scan session investigating the effect of rTMS-augmentation on hypnosis and hypnotizability (120 min scan session) and the second scan session focused on the effect of rTMS-augmented hypnotic analgesia (120 min scan session).

* During the course of the study and upon consultation with the manufacturer, sham setting intensity was lowered to reduce the risk adverse events (e.g., scalp damage).

The study will require that participants participate in an in-person screening visit, a screening MRI scan and 2 MRI scan sessions that include the TMS and hypnosis.

Experimental design. Before each MRI scan session, participants will undergo a preparation session, where hypnotizability and either psychological testing or experimental pain training will be conducted. Volunteer subjects will then participate in 2 MRI scan sessions on two separate days, each lasting approximately 120 mins.

Hypnosis induction procedures. Hypnosis will be induced while the subject is in the scanner though the use of headphones and a pre-recorded induction script. Hypnotic instructions will be standardized, and will involve a simple induction instruction used in our prior research on the brain signature of the hypnotic state and in clinical care. The ability to enter and maintain the hypnotic state through such an induction mechanism in the fMRI environment has been previously demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill 2010 Fibromyalgia Diagnostic Criteria
* Age 18 - 70
* Right-handed
* Agree to and able to have two fMRI scans as well as rTMS sessions
* Willingness to suspend use of analgesic drugs or cough suppressants for 24 hours prior to the scans
* Willingness to suspend us of antidepressant drugs for 2 weeks prior to the scans (6 weeks for fluoxetine)
* Proficiency in English sufficient to complete questionnaires/follow instructions during fMRI assessments
* US Citizen or resident able to receive payment legally
* Low-Moderate Hypnotizability in the Hypnotic Induction Profile (score of 0-8)
* Normal color vision
* Women of childbearing potential must agree to use adequate contraception prior to study entry and continue this for the duration of the study

Exclusion Criteria:

* A medical condition that would contraindicate the use of rTMS
* Any condition that would contraindicate MRI (like ferromagnetic metal in the body)
* Pregnancy or breast feeding
* Any significant neurologic disease, including dementia, multi-infarct dementia, Parkinson's or Huntington's disease, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of significant head trauma
* Current antidepressant use (must be washed out for two weeks prior to starting protocol)
* Inability to stop taking medication contraindicated with treatment
* High Hypnotizability in the Hypnotic Induction Profile (score >8)
* Any significant psychiatric disorder as identified on the Mini Mental State Exam (Dysthymia not an exclusion criteria)
* Color blindness
* Any significant psychiatric disorder as identified on the Mini International Neuropsychiatric Interview
* Previous exposure to rTMS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cojan Y, Piguet C, Vuilleumier P. What makes your brain suggestible? Hypnotizability is associated with differential brain activity during attention outside hypnosis. Neuroimage. 2015 Aug 15;117:367-74. doi: 10.1016/j.neuroimage.2015.05.076. Epub 2015 Jun 3. PMID 26049149
- [Background] Jiang H, White MP, Greicius MD, Waelde LC, Spiegel D. Brain Activity and Functional Connectivity Associated with Hypnosis. Cereb Cortex. 2017 Aug 1;27(8):4083-4093. doi: 10.1093/cercor/bhw220. PMID 27469596
- [Background] Raz A, Fan J, Posner MI. Hypnotic suggestion reduces conflict in the human brain. Proc Natl Acad Sci U S A. 2005 Jul 12;102(28):9978-83. doi: 10.1073/pnas.0503064102. Epub 2005 Jun 30. PMID 15994228
- [Background] Raz A, Shapiro T, Fan J, Posner MI. Hypnotic suggestion and the modulation of Stroop interference. Arch Gen Psychiatry. 2002 Dec;59(12):1155-61. doi: 10.1001/archpsyc.59.12.1155. PMID 12470132
- [Background] Rainville P, Carrier B, Hofbauer RK, Bushnell CM, Duncan GH. Dissociation of sensory and affective dimensions of pain using hypnotic modulation. Pain. 1999 Aug;82(2):159-171. doi: 10.1016/S0304-3959(99)00048-2. PMID 10467921
- [Background] Rainville P, Duncan GH, Price DD, Carrier B, Bushnell MC. Pain affect encoded in human anterior cingulate but not somatosensory cortex. Science. 1997 Aug 15;277(5328):968-71. doi: 10.1126/science.277.5328.968. PMID 9252330
- [Background] Burgmer M, Pogatzki-Zahn E, Gaubitz M, Stuber C, Wessoleck E, Heuft G, Pfleiderer B. Fibromyalgia unique temporal brain activation during experimental pain: a controlled fMRI Study. J Neural Transm (Vienna). 2010 Jan;117(1):123-31. doi: 10.1007/s00702-009-0339-1. Epub 2009 Nov 25. PMID 19937376
- [Background] Short BE, Borckardt JJ, Anderson BS, Frohman H, Beam W, Reeves ST, George MS. Ten sessions of adjunctive left prefrontal rTMS significantly reduces fibromyalgia pain: a randomized, controlled pilot study. Pain. 2011 Nov;152(11):2477-2484. doi: 10.1016/j.pain.2011.05.033. Epub 2011 Jul 20. PMID 21764215
- [Background] Wik G, Fischer H, Bragee B, Finer B, Fredrikson M. Functional anatomy of hypnotic analgesia: a PET study of patients with fibromyalgia. Eur J Pain. 1999 Mar;3(1):7-12. doi: 10.1053/eujp.1998.0093. PMID 10700332
- [Background] Derbyshire SW, Whalley MG, Oakley DA. Fibromyalgia pain and its modulation by hypnotic and non-hypnotic suggestion: an fMRI analysis. Eur J Pain. 2009 May;13(5):542-50. doi: 10.1016/j.ejpain.2008.06.010. Epub 2008 Jul 23. PMID 18653363
- [Background] Orosz A, Jann K, Wirth M, Wiest R, Dierks T, Federspiel A. Theta burst TMS increases cerebral blood flow in the primary motor cortex during motor performance as assessed by arterial spin labeling (ASL). Neuroimage. 2012 Jul 2;61(3):599-605. doi: 10.1016/j.neuroimage.2012.03.084. Epub 2012 Apr 12. PMID 22613775
- [Background] Nettekoven C, Volz LJ, Kutscha M, Pool EM, Rehme AK, Eickhoff SB, Fink GR, Grefkes C. Dose-dependent effects of theta burst rTMS on cortical excitability and resting-state connectivity of the human motor system. J Neurosci. 2014 May 14;34(20):6849-59. doi: 10.1523/JNEUROSCI.4993-13.2014. PMID 24828639
- [Background] Poreisz C, Csifcsak G, Antal A, Levold M, Hillers F, Paulus W. Theta burst stimulation of the motor cortex reduces laser-evoked pain perception. Neuroreport. 2008 Jan 22;19(2):193-6. doi: 10.1097/WNR.0b013e3282f45498. PMID 18185107
- [Background] Goldsworthy MR, Pitcher JB, Ridding MC. Neuroplastic modulation of inhibitory motor cortical networks by spaced theta burst stimulation protocols. Brain Stimul. 2013 May;6(3):340-5. doi: 10.1016/j.brs.2012.06.005. Epub 2012 Jul 5. PMID 22835528
- [Background] Goldsworthy MR, Pitcher JB, Ridding MC. Spaced Noninvasive Brain Stimulation: Prospects for Inducing Long-Lasting Human Cortical Plasticity. Neurorehabil Neural Repair. 2015 Sep;29(8):714-21. doi: 10.1177/1545968314562649. Epub 2014 Dec 11. PMID 25505220
- [Background] Hoeft F, Gabrieli JD, Whitfield-Gabrieli S, Haas BW, Bammer R, Menon V, Spiegel D. Functional brain basis of hypnotizability. Arch Gen Psychiatry. 2012 Oct;69(10):1064-72. doi: 10.1001/archgenpsychiatry.2011.2190. PMID 23026956

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1,058 individuals completed the online interest survey; 157 completed in-person screening, and 101 were randomized to a study arm.
Groups:
- Active rTMS: The active group received active repetitive Transcranial Magnetic Stimulation
  Active repetitive Transcranial Magnetic Stimulation: The investigators performed two applications of 40s of continuous theta-burst stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left dorsolateral prefrontal cortex (DLPFC) was determined by Localite Neuronavigation and targeted at the posterior middle frontal gyrus. The baseline structural scan obtained during the scan 1 was utilized for this localization process. rTMS was delivered using a MagPro TMS system (MagVenture, Denmark).
- Sham rTMS: The sham repetitive Transcranial Magnetic Stimulation group had the stimulation blocked.
  Sham repetitive Transcranial Magnetic Stimulation: This was identical to active rTMS except the stimulation was blocked. Both active and sham repetitive Transcranial Magnetic Stimulation received simulation from a specially designed coil which is capable of delivering either active rTMS or sham rTMS in a manner, which is randomized by the system itself and therefore blinded to the treater. Sham rTMS was delivered using a MagPro TMS system (MagVenture, Denmark).
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 49 | 52
Received Intervention | 40 | 40
Completed Pain Evaluation Study Day | 41 | 44
Completed Mechanistic Evaluation Study Day | 40 | 40
Completed | 40 | 40
Not Completed | 9 | 12
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Severe anxiety | 0 | 1
Not completed — Positive toxicology screen | 0 | 2
Not completed — Claustrophobia | 2 | 2
Not completed — Non-compliance | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active rTMS: The active group received active repetitive Transcranial Magnetic Stimulation
  Active repetitive Transcranial Magnetic Stimulation: The investigators performed two applications of 40s of continuous theta-burst stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left DLPFC was determined by Localite Neuronavigation and targeted at the posterior middle frontal gyrus. The baseline structural scan obtained during the scan 1 was utilized for this localization process. rTMS was delivered using a MagPro TMS system (MagVenture, Denmark).
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 49 | 52 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 47 | 50 | 97
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.8) | 50 (11.6) | 49.47 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 40 | 75
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 49 | 52 | 101

OUTCOME MEASURES:

1. Primary Outcome: The Change in Functional Connectivity (FC) Between the Left Dorsolateral Prefrontal Cortex (L-DLPFC) and the Dorsal Anterior Cingulate Cortex (dACC)
Description: Functional MRI (fMRI) measures changes in oxygenated blood in the brain; at rest these levels fluctuate over time. These fluctuations can be similar between different brain regions. FC is the similarity in fluctuations of these fMRI signals and suggests how strongly two regions communicate with each other. We measured how inhibitory continuous theta-burst stimulation (cTBS) over L-DLPFC changes FC between L-DLPFC and dACC. This was done by estimating z-transformed correlation coefficients (CC) for each voxel (-1 to 1) between the L-DLPFC and dACC pre and post cTBS intervention. Negative FC was assigned to voxels with a weight < 0, positive FC to voxels with weight> 0. Total FC includes positive and negative voxels. The change in FC is regarded as the change in the sum of these weighted voxels from pre to post cTBS for total, positive and negative FC, respectively. Greater sums of voxels correspond to more significant levels of coordinated activity (positive, negative, or total).
Time Frame: Baseline and at 15-20 min post-TMS (up to 30 min)
Population: Participants with resting-state scans for both pre and post-TMS conditions that passed QC and motion-based scan inclusion criteria; outlier data were excluded.
Measure: Mean (Standard Error); unit: Z-transformed CC
Groups:
- Active rTMS: The active group received active repetitive Transcranial Magnetic Stimulation
  Active repetitive Transcranial Magnetic Stimulation: The investigators performed two applications of 40s of continuous theta-burst stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left DLPFC was determined by Localite Neuronavigation and targeted at the posterior middle frontal gyrus. The baseline structural scan obtained during the scan 1 was utilized for this localization process. rTMS was delivered using a MagPro TMS system (MagVenture, Denmark).utilized for this localization process. rTMS will be delivered using a MagPro TMS system (MagVenture, Denmark).
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 26 | 30
Z-transformed CC
  Change in sum of positive z-transformed CC. | 61.98 (21.63) | 4.16 (16.43)
  Change in sum of negative z-transformed CC. | -21.41 (16.8) | -13.22 (16.8)
  Change in sum of all z-transformed CC. | 40.56 (32.34) | -9.06 (28.25)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Examining the Change in sum of positive z-transformed CC; Test type: Superiority; p = 0.035, t-test, 2 sided; 2-sample t-test
Statistical Analysis 2: Comparison: Active rTMS vs Sham rTMS; Examining the change in sum of all z-transformed CC; Test type: Superiority; p = 0.7, t-test, 2 sided — 2-sample t-test
Statistical Analysis 3: Comparison: Active rTMS vs Sham rTMS; Examining the change in sum of negative z-transformed CC; Test type: Superiority — 2-sample t-test; p = 0.11, t-test, 2 sided
Statistical Analysis 4: Comparison: Active rTMS; Examining the change in positive functional connectivity between the L-DLPFC and the dACC within the active group from pre to post TMS; Test type: Superiority; p = 0.008, t-test, 2 sided; One sample(paired) t-test; Mean Difference (Net) = 61.98

2. Secondary Outcome: The Change in the Neural Network Underlying Hypnotic Intensity
Description: Blood oxygen level dependent (BOLD) signal and interleaved TMS-BOLD analyses will be used to determine the effect of active, inhibitory rTMS (cTBS) over L-DLPFC on modulating the neural network that underlies hypnotic intensity.
Time Frame: Baseline and 2 hours
Population: During the study, data were not collected using interleaved TMS-BOLD, as originally planned.
Groups:
- Active rTMS: The active group received active repetitive Transcranial Magnetic Stimulation.
  Active repetitive Transcranial Magnetic Stimulation: The investigators performed two applications of 40s of continuous theta-burst stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left DLPFC was determined by Localite Neuronavigation and targeted at the posterior middle frontal gyrus. The baseline structural scan obtained during the scan 1 was utilized for this localization process. rTMS was delivered using a MagPro TMS system (MagVenture, Denmark).
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Hypnotic Induction Profile Score
Description: The investigators used the Hypnotic Induction Profile (HIP) to determine the effect of active, inhibitory rTMS (cTBS) over L-DLPFC on enhancing hypnotizability.
  HIP scores range from 0 to 10 (low to high hypnotizability).
Time Frame: Baseline and Immediately post rTMS (up to 30 min)
Population: Participants with available data are included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 40 | 40
score on a scale | .63 (1.18) | .31 (1.67)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Non-parametric analysis, comparison of change (post-treatment minus pre-treatment); Test type: Other; p = 0.046, Mann-Whitney U-test 2-tailed; Mann-Whitney U statistic = 601
Statistical Analysis 2: Comparison: Active rTMS vs Sham rTMS; Non-parametric analysis, comparison of change (post-treatment minus pre-treatment); Test type: Other; Cohen's R = 0.25 — Estimate of effect size

4. Secondary Outcome: Change in The Hypnosis Intensity Scale
Description: The investigators used the Hypnotic Intensity Scale (HIS) to determine the effect of active, inhibitory rTMS (cTBS) over L-DLPFC on enhancing hypnotic intensity.
  HIS scores range from 0 to 10 (low to high hypnotic intensity).
Time Frame: Baseline and immediately post rTMS (up to 2 hrs)
Population: Participants who completed the protocol and completed HIS ratings are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 40 | 39
score on a scale | .475 (2.242) | -.128 (1.490)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Pre- to post-rTMS change in HIS scores were calculated for both Active and Sham conditions. Two-tailed t-tests were used to evaluate the difference between the two conditions' change scores; Test type: Superiority — We assessed the superiority of active over sham; p = .412, Mann-Whitney U-test 2-tailed; Mann-Whitney U statistic = 702.5

5. Secondary Outcome: The Change in Functional Connectivity (FC) Within The Neural Network Underlying Conflict Regulation.
Description: We examined the effect of active, inhibitory cTBS over L-DLPFC on functional connectivity (FC) in key nodes in the neural network underlying the conflict regulation system. FC between each voxel in the L-DLPFC and the entire dACC was established by estimating z-transformed correlation coefficients (CC) for each voxel (-1 to 1) pre and post cTBS intervention. This paradigm was also used for voxels in the Default Mode Network (DMN) (Schaefer, 2018; Yeo, 2011) to the entire right inferior frontal gyrus (rIFG). Negative FC was assigned to voxels with a weight < 0, positive FC to voxels with weight > 0. Total FC includes positive and negative voxels. The change in FC is regarded as the change in the sum of these weighted voxels from pre to post cTBS for total, positive and negative FC, respectively. Greater sums of voxels correspond to more significant levels of coordinated activity (positive, negative, or total).
Time Frame: Baseline and at 15-20 min post-TMS (up to 30 min)
Population: Population consisted of patients with fibromyalgia who underwent either active or sham cTBS either in combination with hypnosis or without it. Participants were excluded from the original sample for 1) fMRI imaging problems, 2) missing data. For the analyses below additional outliers were excluded on a test by test basis.
Measure: Mean (Standard Deviation); unit: Z-transformed CC
Groups:
- Active rTMS: The active group will receive repetitive Transcranial Magnetic Stimulation
  repetitive Transcranial Magnetic Stimulation: The investigators will perform two applications of 40s of continuous theta-burst stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left DLPFC will be determined by Localite Neuronavigation and targeted at the posterior middle frontal gyrus. The baseline structural scan obtained during the scan 1 will be utilized for this localization process. rTMS will be delivered using a MagPro TMS system (MagVenture, Denmark).
- Sham rTMS: The sham repetitive Transcranial Magnetic Stimulation group will have the stimulation blocked.
  Sham repetitive Transcranial Magnetic Stimulation: This will be identical to active rTMS except the stimulation will be blocked. Both active and sham repetitive Transcranial Magnetic Stimulation will receive simulation from a specially designed coil which is capable of delivering either active rTMS or sham rTMS in a manner, which is randomized by the system itself and therefore blinded to the treater. rTMS will be delivered using a MagPro TMS system (MagVenture, Denmark).
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 25 | 24
Z-transformed CC
  Change in sum of all z-transformed CC in L-DLPFC.: number analyzed (Participants) | 23 | 23
  Change in sum of all z-transformed CC in L-DLPFC. | 0.01 (0.14) | -0.003 (0.13)
  Change in sum of positive z-transformed CC in L-DLPFC.: number analyzed (Participants) | 23 | 23
  Change in sum of positive z-transformed CC in L-DLPFC. | 33.76 (136.5) | 6.39 (99.82)
  Change in sum of negative z-transformed CC in L-DLPFC.: number analyzed (Participants) | 23 | 23
  Change in sum of negative z-transformed CC in L-DLPFC. | -20.36 (88.88) | -10.11 (96.55)
  Change in sum of all z-transformed CC in DMN.: number analyzed (Participants) | 23 | 23
  Change in sum of all z-transformed CC in DMN. | 0.004 (0.05) | -0.01 (0.05)
  Change in sum of positive z-transformed CC in DMN.: number analyzed (Participants) | 23 | 23
  Change in sum of positive z-transformed CC in DMN. | -31.20 (137.73) | 21.12 (153.54)
  Change in sum of negative z-transformed CC in DMN.: number analyzed (Participants) | 23 | 23
  Change in sum of negative z-transformed CC in DMN. | 51.35 (243.68) | -67.65 (219.05)

6. Secondary Outcome: The Change in Stroop Performance
Description: Stroop effect is measured by the response time of a participant during the stroop task. Increases in response time indicate increased stroop effect (SE) and vice versa.
Time Frame: Baseline and at 15-20 min post-TMS (up to 30 min)
Population: Population consisted of patients with fibromyalgia who underwent either active or sham cTBS either in combination with hypnosis or without it. Participants were excluded from the original sample for 1) poor Stroop task performance, 2) fMRI imaging problems, 3) missing data. For the analyses below additional outliers were excluded on a test by test basis.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 23 | 24
Seconds
  Mean difference in change in Stroop effect (s) without hypnosis (TMS - no TMS) condition. | 0.01 (0.1) | -0.02 (0.082)
  Mean difference in change in Stroop effect (s) with hypnosis (TMS - no TMS) condition.: number analyzed (Participants) | 23 | 23
  Mean difference in change in Stroop effect (s) with hypnosis (TMS - no TMS) condition. | -0.04 (0.12) | -0.009 (.10)

7. Secondary Outcome: Stroop Task
Description: Active, inhibitory cTBS effect over L-DLPFC on the neural network that underlies the hypnotic Stroop modulation effect was determined by first estimating the average of connectivity weights for all parcel pairs linking Ventral Attentional Network (VAN) to the DMN. Parcels are determined by extracting mean resting state BOLD time-series for each region of the Schaefer 100 parcellation. A correlation matrix between all parcels is created and FC weights for each pair are established by estimating z-transformed correlation coefficients (CC) (-1 to 1). Each parcel pair is then assigned to one of the 7 resting state networks defined by Yeo et al., (2011). Negative FC is defined for parcel pairs with a weight < 0, positive FC pairs with weight > 0 and total FC includes all pairs. FC is thus the average value between parcel pairs in the DMN and VAN pre/post TMS. Greater sums of weighted pairs correspond to more significant levels of coordinated activity (positive, negative, or total).
Time Frame: Baseline and at 15-20 min post-TMS (up to 30 min)
Population: Subjects who had pre and post TMS resting-state fMRI scans that passed QC and motion-based inclusion criteria
Measure: Mean (Standard Error); unit: Z-transformed CC
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 27 | 30
Z-transformed CC | -0.026 (0.0265) | 0.155 (0.0297)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Test type: Superiority; p = 0.037, t-test, 2 sided; 2-sample t-test
Statistical Analysis 2: Comparison: Active rTMS; Test type: Superiority; p = 0.063, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham rTMS; Test type: Superiority; p = 0.31, t-test, 2 sided

8. Secondary Outcome: Linear Relationship Between the Change in FC of the VAN to the DMN and the Change in Stroop Performance (Correlation Coefficient) With no Hypnosis Intervention.
Description: Spearman's correlation was used to determine the linear relationship between the response time taken to answer incongruent Stroop task blocks (a measure of Stroop performance) and the change the resting-state network FC between the VAN and the DMN when no hypnosis intervention was implemented.
Time Frame: Baseline and at 15-20 min post-TMS (up to 1 hr)
Population: Population consisted of patients with fibromyalgia who underwent either active or sham cTBS either in combination with hypnosis or without it. Participants were excluded from the original sample for 1) poor Stroop task performance, 2) fMRI imaging problems, 3) missing data. Subjects who had pre and post TMS resting-state fMRI scans that passed QC and motion-based inclusion criteria were included.
Measure: Number; unit: Correlation Coefficient
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 27 | 30
Correlation Coefficient | 0.18 | -0.58

9. Secondary Outcome: Linear Relationship Between the Change in FC of the VAN to the DMN and the Change in Stroop Performance (Correlation Coefficient) With Hypnosis Intervention.
Description: Spearman's correlation was used to determine the linear relationship between the response time taken to answer incongruent Stroop task blocks (a measure of Stroop performance) and the change the resting-state network FC between the VAN and the DMN when the hypnosis intervention was implemented.
Time Frame: Baseline and at 15-20 min post-TMS (up to 1 hr)
Population: as for outcome 8
Measure: Number; unit: Correlation Coefficient
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 27 | 30
Correlation Coefficient | 0.16 | 0.16

10. Secondary Outcome: Linear Relationship Between the Change in FC of the VAN to the DMN and the Change in Stroop Interference (Correlation Coefficient) With no Hypnosis Intervention.
Description: Spearman's correlation was used to determine the linear relationship between the Stroop interference and the change the resting-state network FC between the VAN and the DMN when no hypnosis intervention was implemented.
  In psychology, the Stroop effect is the delay in reaction time between congruent and incongruent stimuli.
Time Frame: Baseline and at 15-20 min post-TMS (up to 1 hr)
Population: as for outcome 8
Measure: Number; unit: Correlation Coefficient
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 27 | 30
Correlation Coefficient | 0.24 | -0.44

11. Secondary Outcome: Linear Relationship Between the Change in FC of the VAN to the DMN and the Change in Stroop Interference (Correlation Coefficient) With Hypnosis Intervention.
Description: Spearman's correlation was used to determine the linear relationship between the Stroop interference and the change the resting-state network FC between the VAN and the DMN when the hypnosis intervention was implemented.
  In psychology, the Stroop effect is the delay in reaction time between congruent and incongruent stimuli.
Time Frame: Baseline and at 15-20 min post-TMS (up to 1 hr)
Population: as for outcome 8
Measure: Number; unit: Correlation Coefficient
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 27 | 30
Correlation Coefficient | 0.07 | 0.28

12. Secondary Outcome: Change in the Numeric Pain Rating Scale
Description: To determine the effect of active, inhibitory rTMS (cTBS) over L-DLPFC on modulating the neural network that underlies hypnotic analgesia (HA).
  Numeric Pain Rating Scale scores range from 0 to 10 (low to high pain intensity).
Time Frame: Baseline and immediately post-rTMS (up to 30 minutes)
Population: Participants with available data are included in the analysis
Measure: Mean (Standard Error); unit: mean change of scores on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 38 | 42
mean change of scores on a scale
  Non-hypnosis condition | -0.13 (0.20) | 0.19 (0.19)
  Hypnosis condition | -0.09 (0.20) | -0.05 (0.19)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; We used standard mixed-effects modeling to estimate the change (slope) in pain in our 2*2 pre- and post-assessment design. Pain ratings were calculated by averaging pain ratings across 5 assessments under four conditions (TMS with hypnosis, TMS without hypnosis, Sham with hypnosis, Sham without hypnosis). Based on these change estimates, we derived the two main effects (TMS, Hypnosis) and their interaction effect on the change in pain from the pre- to post-treatment assessment; Test type: Superiority — We assessed the superiority of active over sham; p = 0.49, Mixed-effects model; Cohen's d = -0.234

13. Secondary Outcome: Change in Sense of Agency Rating Scale (SOARS)
Description: The investigators used the Sense of Agency Rating Scale (SOARS) to determine the effect of active, inhibitory rTMS (cTBS) over L-DLPFC on altering the subjective sense of agency during hypnotizability.
  SOARS scores are calculated for Involuntariness and Effortlessness, each range from 0 to 35 (low to high).
Time Frame: Baseline and immediately post-rTMS (up to 30 min)
Population: Participants who completed the protocol and completed all items of the SOARS are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 35 | 33
score on a scale
  Involuntariness | .3529 (3.3654) | 1.1034 (3.8391)
  Effortlessness | .8857 (3.5378) | .2727 (3.1551)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Pre- to post-rTMS change in SOARS scores were calculated for both Active and Sham conditions. Two-tailed t-tests were used to evaluate the difference between the two conditions' change scores; Test type: Superiority — We assessed the superiority of active over sham; p = .454, t-test, 2 sided

14. Secondary Outcome: Metabolic Alterations in Fibromyalgia (FMS) Defined by Excitatory / Inhibitory Ratio
Description: E/I ratio is defined as the logarithm of the concentration of Glx (excitatory neurotransmitter metabolite complex) /GABA+ (inhibitory neurotransmitter metabolite complex) relative to either water or creatine peak signal and it is a unitless measure ranging from -1 to 1. Logarithmic transformations are used to account for non-normal distributions of metabolite concentrations across participants and ratios > 0 are thought to be excitatory neurotransmitter dominant while ratios <0 are thought to be inhibition dominant.
Time Frame: Baseline Scan (up to 15 min)
Population: Participants with baseline MegaPress scan data
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Baseline Fibromyalgia MRSPEC Analysis: MEGA-PRESS (Mescher M, Merkle H, Kirsch J, Garwood M, Gruetter R, 1998) Spectra were acquired during baseline scanning for TMS-naive participants with Fibromyalgia before any intervention as part of an F32 grant.
Arm/Group | Baseline Fibromyalgia MRSPEC Analysis
Number analyzed (Participants) | 51
Ratio
  GABA+/Cr | 0.10 (0.02)
  GABA+/Water | 1.72 (0.33)
  Glx/Cr | 0.09 (0.01)
  Glx/Water | 5.43 (0.82)
  Log E/I Cr | -0.06 (0.08)
  Log E/I Water | 0.50 (0.08)
Statistical Analysis 1: Comparison: Baseline Fibromyalgia MRSPEC Analysis; In people with FMS, the linear relationship between Thermal Pain Tolerance and E/I ratio as it relates to water was assessed; Test type: Other — Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to water and Thermal Pain Tolerance with E/I as the independent variable and Thermal Pain Tolerance as the dependent variable; p = 0.023, Regression, Linear; (R² = .104, F(2,48) = 2.794, β = .320, p = .023)
Statistical Analysis 2: Comparison: Baseline Fibromyalgia MRSPEC Analysis; In people with FMS, the linear relationship between Thermal Pain Threshold and E/I ratio as it relates to water was assessed; Test type: Other — Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to water and Thermal Pain Threshold with E/I as the independent variable and Thermal Pain Threshold as the dependent variable; p = 0.043, Regression, Linear; (R² = .081, F(1,49) = 4.315, β = .284, p = .043)
Statistical Analysis 3: Comparison: Baseline Fibromyalgia MRSPEC Analysis; In people with FMS, the linear relationship between Thermal Pain Tolerance and E/I ratio as it relates to creatine was assessed; Test type: Other — Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to creatine and Thermal Pain Tolerance with E/I as the independent variable and Thermal Pain Tolerance as the dependent variable; p = 0.022, Regression, Linear; (R² = .103, F(1,49) = 5.632, β = .321, p = .022)
Statistical Analysis 4: Comparison: Baseline Fibromyalgia MRSPEC Analysis; In people with FMS, the linear relationship between Thermal Pain Threshold and E/I ratio as it relates to creatine was assessed; Test type: Other — Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to creatine and Thermal Pain Threshold with E/I as the independent variable and Thermal Pain Threshold as the dependent variable; p = 0.041, Regression, Linear; (R² = .083, F(1,49) = 4.425, β = .288, p = .041)

15. Secondary Outcome: Alterations in Pain Perception in Fibromyalgia
Description: To characterize clinical pain measures, which are defined as thermal pain threshold and thermal pain tolerance. Thermal pain threshold is determined as the temperature of a thermode determined as painful (degrees Celsius) by a participant. Thermal pain tolerance extends this to the point at which discontinuation is necessary (degrees Celsius).
Time Frame: Baseline visit (up to 30 min)
Population: Participants with baseline MegaPress scan data
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Baseline Fibromyalgia MRSPEC Analysis
Number analyzed (Participants) | 51
Degrees Celsius
  Thermal Pain Tolerance (degrees Celsius) | 47.8 (2.51)
  Thermal Pain Threshold (degrees Celsius) | 44.6 (3.55)

16. Secondary Outcome: Linear Regression of Thermal Pain Threshold to Logarithm of E/I Ratio as it Relates to Water in Fibromyalgia (Coefficient of Determination)
Description: Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to water and Thermal Pain Threshold with E/I as the independent variable and Thermal Pain Threshold as the dependent variable.
Time Frame: Baseline visit (up to 45 min)
Population: Participants with baseline MegaPress scan data
Measure: Number; unit: Coefficient of determination
Arm/Group | Baseline Fibromyalgia MRSPEC Analysis
Number analyzed (Participants) | 51
Coefficient of determination | 0.104

17. Secondary Outcome: Linear Regression of Thermal Pain Tolerance to Logarithm of E/I Ratio as it Relates to Water in Fibromyalgia (Coefficient of Determination)
Description: Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to water and Thermal Pain Tolerance with E/I as the independent variable and Thermal Pain Tolerance as the dependent variable.
Time Frame: Baseline visit (up to 45 min)
Population: Participants with baseline MegaPress scan data
Measure: Number; unit: Coefficient of determination
Arm/Group | Baseline Fibromyalgia MRSPEC Analysis
Number analyzed (Participants) | 51
Coefficient of determination | 0.104

18. Secondary Outcome: Linear Regression of Thermal Pain Threshold to Logarithm of E/I Ratio as it Relates to Creatine in Fibromyalgia (Coefficient of Determination)
Description: Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to creatine and Thermal Pain Threshold with E/I as the independent variable and Thermal Pain Threshold as the dependent variable.
Time Frame: Baseline visit (up to 45 min)
Population: Participants with baseline MegaPress scan data
Measure: Number; unit: Coefficient of determination
Arm/Group | Baseline Fibromyalgia MRSPEC Analysis
Number analyzed (Participants) | 51
Coefficient of determination | 0.083

19. Secondary Outcome: Linear Regression of Thermal Pain Tolerance to Logarithm of E/I Ratio as it Relates to Creatine in Fibromyalgia (Coefficient of Determination)
Description: Linear regression was used to evaluate the scalar relationship between E/I ratio as it relates to creatine and Thermal Pain Tolerance with E/I as the independent variable and Thermal Pain Tolerance as the dependent variable.
Time Frame: Baseline visit (up to 45 min)
Population: Participants with baseline MegaPress scan data
Measure: Number; unit: Coefficient of determination
Arm/Group | Baseline Fibromyalgia MRSPEC Analysis
Number analyzed (Participants) | 51
Coefficient of determination | 0.103

20. Secondary Outcome: Metabolic Changes in L-DLPFC Pre- and Post-rTMS
Description: To determine the relationship between the metabolic alterations pre and post-rTMS. Metabolic changes as measured by MEGA-PRESS spectroscopy were assessed by quantification of excitatory (Glx) and inhibitory (GABA+) neurotransmitter complexes. The E/I ratio is defined as the logarithm of the concentration of Glx/GABA+relative to either the reference water or creatine signal and it is a unitless measure ranging from -1 to 1. Logarithmic transformations are used to account for non-normal distributions of metabolite concentrations across participants and ratios > 0 are thought to be excitatory neurotransmitter dominant while ratios <0 are thought to be inhibition dominant.
Time Frame: Baseline Scan and at 15-20 min post-TMS (up to 30 min)
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 14 | 21
Ratio
  Log E/I Water Pre-TMS | 0.487 (0.075) | 0.486 (0.092)
  Log E/I Water Post-TMS | 0.494 (0.073) | 0.505 (0.109)
  Log E/I Creatine Pre-TMS | -0.075 (0.075) | -0.076 (0.092)
  Log E/I Creatine Post-TMS | -0.068 (0.073) | -0.057 (0.108)
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Standard ANCOVA testing whether the Post-TMS E/I relative to creatine is predicted for each subject by the intervention (Active / Sham) while covarying for the Pre-TMS E/I ratio relative to creatine; Test type: Superiority; p = 0.728, ANCOVA
Statistical Analysis 2: Comparison: Active rTMS vs Sham rTMS; Standard ANCOVA testing whether the Post-TMS E/I relative to water is predicted for each subject by the intervention (Active / Sham) while covarying for the Pre-TMS E/I ratio relative to water; Test type: Superiority; p = 0.720, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/52
Other Adverse Events (participants affected / at risk) | 1/49 | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=49) | Sham rTMS (N=52)
Medication Withdrawal During Washout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — One patient experienced medication withdrawal during the washout period for the study.
Headache / Scalp Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One Participant experienced a headache and scalp irritation under the site of the TMS coil (a common side effect) during active treatment.
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Dizziness from MRI machine during scanning session

LIMITATIONS AND CAVEATS:
fMRI BOLD data were preprocessed using fMRIPrep 1.5.10 (Esteban, Markiewicz, et al. (2018); Esteban, Blair, et al. (2018); RRID:SCR_016216), which is based on Nipype 1.4.2 (Gorgolewski et al. (2011); Gorgolewski et al. (2018); RRID:SCR_002502) with MNI152NLin2009cAsym and anatomical output spaces. BOLD time series were bandpass filtered to include data in the window of 0.0025-0.025 Hz, which is on the low end of the spectrum. A more typical bandpass window is 0.01 - 0.1 Hz.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Original Protocol and Statistical Methods (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT02969707/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Revised Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02969707/SAP_003.pdf
  • Informed Consent Form (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02969707/ICF_002.pdf